CLINICAL TRIAL: NCT02466581
Title: A Multicenter, Randomized, Open-label, Blinded-assessor, Follow-up, Phase 4 Study in Patients With Rheumatoid Arthritis Who Have Completed the Initial Treatment Part in the NORD-STAR Study and Have Reached Stable Low Disease Activity
Brief Title: Dose Reduction for Early Rheumatoid Arthritis Patients With Low Disease Activity
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Karolinska Institutet (Other)
Responsible Party: Principal Investigator, Ronald van Vollenhoven, prof., Professor, Karolinska Institutet
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: CO-STAR; 2014-002374-36 (EudraCT Number); 2014/1705-31/3 (Other: Regional Ethical Review Board)
Record Dates: First submitted 2015-05-29; First posted 2015-06-09 (Estimated); Last update posted 2022-07-08 (Actual); Status verified 2022-07

CONDITIONS: Rheumatoid Arthritis
MeSH Terms: conditions — Arthritis, Rheumatoid | interventions — Sulfasalazine; Hydroxychloroquine; Prednisolone; Certolizumab Pegol; Abatacept; tocilizumab

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Arm 1 (Active Comparator): Patients keep the intervention they had in the NORD-STAR-study (NCT01491815), i.e. one of the four below:
  1. Sulphasalazine + Hydroxychloroquine OR Prednisolone plus Methotrexate and steroids
  2. Cimzia plus Methotrexate and steroids
  3. Orencia plus Methotrexate and steroids
  4. RoActemra plus Methotrexate and steroids
  This intervention is de-escalated starting at randomization.
  Interventions: Drug: Sulphasalazine + Hydroxychloroquine OR Prednisolone; Biological: Cimzia; Biological: Orencia; Biological: RoActemra
- Arm 2 (Active Comparator): Patients keep the intervention they had in the NORD-STAR-study (NCT01491815), i.e. one of the four below:
  1. Sulphasalazine + Hydroxychloroquine OR Prednisolone plus Methotrexate and steroids
  2. Cimzia plus Methotrexate and steroids
  3. Orencia plus Methotrexate and steroids
  4. RoActemra plus Methotrexate and steroids
  This intervention is de-escalated starting 24 weeks after randomization.
  Interventions: Drug: Sulphasalazine + Hydroxychloroquine OR Prednisolone; Biological: Cimzia; Biological: Orencia; Biological: RoActemra

INTERVENTIONS:
Drug: Sulphasalazine + Hydroxychloroquine OR Prednisolone — Methotrexate: 25mg/week. SSZ: 2 g/day. HCQ: 35 mg/kg/week (Finland and Denmark) Methotrexate: 25mg/week. Prednisolone 20 mg/day tapered in 9 weeks to 5 mg/day, discontinued after 9 months. (Sweden, Norway, and Iceland)
  Other Names: SSZ+HCQ or Prednisolone
Biological: Cimzia — Certolizumab-pegol: 200 mg s.c. every other week. Methotrexate: 25mg/week
  Other Names: Certolizumab-pegol
Biological: Orencia — Abatacept: 125 mg s.c. every week. Methotrexate: 25mg/week
  Other Names: Abatacept
Biological: RoActemra — Tocilizumab is given as 4-weekly infusions at dosage 8 mg/kg or 162 mg in solution s.c. every week. Methotrexate: 25mg/week
  Other Names: Tocilizumab

SUMMARY:
This is an international (Nordic) trial designed to compare the safety and efficacy of active conventional therapy (ACT) and three biologic treatments (Certolizumab-pegol, Abatacept or Tocilizumab) in subjects with early rheumatoid arthritis (RA). The global aim of this study is to assess and compare two alternative de-escalation strategies in patients who achieved low disease activity during first-line therapy in the NORD-STAR study.

DETAILED DESCRIPTION:
25 patients have been included in the study of which 1 has had an early termination an 22 have completed the full study.

ELIGIBILITY:
Inclusion Criteria:

1. Subject has been enrolled in the NORD-STAR study according to that study inclusion criteria (and did not meet any of the exclusion criteria in that study).
2. Subject has low-disease-activity according to: 2.8 < CDAI ≤ 10.0, from week 56 in the NORD-STAR study, i.e. during 24 weeks before randomization.
3. Subject has not more than 3 tender out of the 28 joints.
4. According to the investigators opinion the remaining findings are not due to significant active disease (RA).
5. Female subject is either not of childbearing potential (postmenopausal, surgically sterile etc.), or is of childbearing potential and practicing one of the following methods of birth control throughout the study and for 150 days after study completion:

   * Intrauterine device (IUD)
   * Contraceptives (oral, parenteral, patch) for three months prior to study drug administration)
   * A vasectomized partner
6. Subject is judged to be in good general health as determined by the principal investigator.
7. Subject must be able and willing to provide written informed consent and comply with the requirements of this study protocol.

Exclusion Criteria:

1. Subject has left the NORD-STAR study due to moderate or high disease activity (CDAI ≥ 10.0) or for other medically important event(s).
2. Patient is eligible for treatment part 2 (A or B) in the NORD-STAR study.
3. Active infection of any kind (excluding fungal infections of nail beds), or any major episode of infection requiring hospitalization within 4 weeks prior to randomization.
4. Subject has a poorly controlled medical condition, such as uncontrolled diabetes, unstable heart disease, congestive heart failure, recent cerebrovascular accidents and any other condition which, in the opinion of the investigator, would put the subject at risk by participation in the study.
5. Subject has a history of clinically significant hematologic (e.g., severe anemia, leukopenia, thrombocytopenia), renal or liver disease (e.g., fibrosis, cirrhosis, hepatitis).
6. Subject has history of neurologic symptoms suggestive of central nervous system (CNS) demyelinating disease and/or diagnosis of central demyelinating disease.
7. Subject has history of cancer or lymphoproliferative disease. Allowable exceptions:

   1. Successfully treated cutaneous squamous cell or basal cell carcinoma
   2. Localized carcinoma in situ of the cervix
   3. Curatively treated malignancy (treatment terminated) > 5 years prior to randomization.
8. Subject has a history of listeriosis, histoplasmosis, untreated TB, persistent chronic infections, or recent active infections requiring hospitalization or treatment with intravenous (i.v.) anti-infectives within 30 days or oral anti-infectives within 14 days prior to randomization.
9. Female subject who is pregnant or breast-feeding or considering becoming pregnant during the study or within 150 days after the last dose of study medication.
10. Men who are planning to father a child during the time they are included in the study.
11. Subject has a history of clinically significant drug or alcohol usage in the last year.
12. Subject has a chronic widespread pain syndrome.
13. Subject is considered by the investigator, for any reason, to be an unsuitable candidate for the study.
14. Subject is unwilling to comply with the study protocol.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 25 (Actual)
Dates: Start 2015-02-03 (Actual); Primary Completion 2023-07-22 (Estimated); Study Completion 2023-12 (Estimated)

PRIMARY OUTCOMES:
Proportion of patients maintaining low disease activity after dose reduction | 24 weeks after dose reduction
  The proportion of patients, with early dose reduction vs late dose reduction, who maintain low disease activity (2.8 < CDAI ≤ 10.0) at the time point 24 weeks after the dose was first reduced.

CONTACTS AND LOCATIONS:
Overall Officials: Ronald van Vollenhoven, MD, Prof., Principal Investigator — Karolinska Institutet
Locations (8):
- Sweden (8):
  - Sahlgrenska University Hospital, Gothenburg
  - The Karolinska University Hospital, Huddinge
  - Linköping University Hospital, Linköping
  - Skåne University Hospital, Lund
  - Skåne University Hospital, Malmo
  - The Karolinska University Hospital, Solna
  - Karolinska Institutet, Stockholm
  - Academic Specialist Center, Stockholm

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Glinatsi D, Heiberg MS, Rudin A, Nordstrom D, Haavardsholm EA, Gudbjornsson B, Ostergaard M, Uhlig T, Grondal G, Horslev-Petersen K, van Vollenhoven R, Hetland ML. Head-to-head comparison of aggressive conventional therapy and three biological treatments and comparison of two de-escalation strategies in patients who respond to treatment: study protocol for a multicenter, randomized, open-label, blinded-assessor, phase 4 study. Trials. 2017 Apr 4;18(1):161. doi: 10.1186/s13063-017-1891-x. PMID 28376912